CLINICAL TRIAL: NCT04381299
Title: Is Autologous Platelet Rich Plasma Able To Restore Ovarian Function? A Prospective Randomized Control Trial.
Brief Title: Will Autologous Platelet Rich Plasma Able To Restore Ovarian Function?
Status: Active, not recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2004-ABU-003-LM
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Infertility; IVF; Premature Ovarian Failure; Anti-Mullerian Hormone Deficiency
MeSH Terms: conditions — Infertility; Primary Ovarian Insufficiency | interventions — Saline Solution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: The cortex of selected ovary will be injected with 1 mL of autologous platelet rich plasma. Up to ten different sites will be injected under ultrasound guidance. In the surgical report, the surgeon will state how many punctures have been done.
  Interventions: Other: autologous platelet rich plasma
- Control: The cortex of contralateral ovary will be injected with 1 mL of saline solution (SS). Up to ten different sites will be injected under ultrasound guidance. In the surgical report, the surgeon will state how many punctures have been done.
  Interventions: Other: saline solution

INTERVENTIONS:
Other: autologous platelet rich plasma — The cortex of selected ovary will be injected with 1 mL of autologous platelet rich plasma. Up to ten different sites will be injected under ultrasound guidance. In the surgical report, the surgeon will state how many punctures have been done.
  Groups: Intervention
Other: saline solution — The cortex of contralateral ovary will be injected with 1 mL of saline solution (SS). Up to ten different sites will be injected under ultrasound guidance. In the surgical report, the surgeon will state how many punctures have been done.
  Groups: Control

SUMMARY:
A-PRP (Autologous Platelet Rich Plasma) is becoming widely used in a variety of medical procedures seeking tissue remodeling and/or healing as an intervention. To date, applications in orthopedics, wound healing, dermatology and plastic surgery have gained general acceptance, primarily as the role of platelets and their activation in tissue repair and recovery has become better understood at a cellular and molecular level. This study will involve adult women with a diagnosis of Premature ovarian insufficiency (POI) willing to perform an IVF/ICSI treatment.

DETAILED DESCRIPTION:
POI is a loss of normal function before age 40, leading to infertility and hypergonadotropic hypoestrogenism. Currently, no optimal regimen exists to ameliorate ovarian function. The options to conceive genetically related offspring, are limited. Typically, affected patients end up with egg donation or adoption as an alternative .

A-PRP is plasma with a concentration of platelets above the blood baseline. A-PRP is developed from autologous blood. Within A-PRP, the concentration of platelets delivers an increased number of growth factors. PRP is becoming widely used in a variety of medical procedures seeking tissue remodeling and/or healing as an intervention. To date, applications in orthopedics, wound healing, dermatology and plastic surgery have gained general acceptance, primarily as the role of platelets and their activation in tissue repair and recovery has become better understood at a cellular and molecular level. This knowledge base provides a foundation for the present study because of the ready availability of FDA-approved kits for autologous PRP preparations and the recognition that the aging ovary acquires tissue pathologies in the form of wound healing and fibrosis as a result of repeat ovulations over the reproductive lifespan of women. Since PRP is an autologous blood product and is widely used via injection into various organs and tissues, safety concerns are minimal.

This study will involve adult women with a diagnosis of Premature ovarian insufficiency (POI) willing to perform an IVF/ICSI treatment. A-PRP will be prepared using Eclipse PRP Kit which is approved by US FDA for preparation of PRP. Consenting participants will receive injections of autologous Platelet Rich Plasma (A-PRP) in one randomly selected ovary under ultrasound guidance performed under IV sedation. As it is suggested that only mechanical stimulation by biopsy/scratch could be a potentially effective method for follicle activation, the other ovary will be injected with the same amount of Saline Solution (SS) as control, to replicate the same mechanical effect. Randomization will determine whether the right or left ovary will be treated. Follow up of the participants will be performed with transvaginal ultrasound and hormonal tests including AMH, FSH, LH, estradiol and progesterone, every 10 days for the next 3 months after the injection. If ovarian activity is detected, the participant will undergo an IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women 40 years of age and younger with documented primary ovarian insufficiency (12).
* Normal Karyotype
* BMI </= 35 kg/m2
* Oligo/amenorrhea for at least 4 months
* FSH > 25 IU/mL
* AMH </= 0,1 ng/ml
* No evidence of follicles > 4mm
* Must have two ovaries of approximately equal volume.
* Willingness to undergo further fertility treatment, including IVF if there is evidence of response
* A transvaginal scan including Doppler for arteria ovarica will be performed previously to the surgical procedure.

Exclusion Criteria:

* Premature ovarian failure due to a genetic origin, such as Turner's Syndrome or chromosomal abnormality.
* Oncological diseases (specially, skeletal system and blood).
* Autoimmune diseases, for example, lupus erythematosus, etc.
* Previous treatments including radiotherapy or chemotherapy.
* Other conditions not suitable for surgical procedures and/or anesthesia.
* Anticoagulant or antiaggregant treatment.
* Acute and chronic infectious diseases.
* Active substance abuse or dependence.
* Major Mental health disorder.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Adult women with primary or secondary infertility with a diagnosis of POI, willing to perform an IVF treatment.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Appearance of new ovarian follicles (number of follicles growing) with evidence of estradiol production. | 12 weeks
  Evaluate the difference of number of follicles growing, means values will be calculated at the two points time (baseline and 12 weeks).
  Means differences will be verified using the t test analysis (after confirming the normal distribution of the data by means of Kolmogorov-Smirnoff tests. If normal distribution is not confirmed a non-parametric anova test will be used. This rule will be applied to all analysis

SECONDARY OUTCOMES:
Increase in serum AMH above the baseline level | 12 weeks
  Evaluate the difference of AMH levels between time, means values will be calculated at the two points time (baseline and 12 weeks). Means differences will be verified using the t test analysis.
Increase in AFC above the baseline level in 12 weeks | 12 weeks
  Evaluate the difference of AFC levels between groups, means values will be calculated at the two points time (baseline and 12 weeks). Means differences will be verified using the t test analysis
Total number of retrieved oocytes in an IVF cycle. | 1 day
  Number of retrieved oocytes will be calculated in the IVF cycle: total and per groups (per ovary)
Pregnancy rates | 40 weeks
  Pregnancy rates:
  1. Biochemical pregnancy rate: Percentage of bHCG above 15 IU/ml per embryo transfer performed.
  2. Clinical pregnancy rate: percentage of pregnancies with fetal heart rate positive per embryo transfer performed. Miscarriage rate: percentage of miscarriages per embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Laura Melado, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ford EA, Beckett EL, Roman SD, McLaughlin EA, Sutherland JM. Advances in human primordial follicle activation and premature ovarian insufficiency. Reproduction. 2020 Jan;159(1):R15-R29. doi: 10.1530/REP-19-0201. PMID 31376814
- [Background] Zhang X, Han T, Yan L, Jiao X, Qin Y, Chen ZJ. Resumption of Ovarian Function After Ovarian Biopsy/Scratch in Patients With Premature Ovarian Insufficiency. Reprod Sci. 2019 Feb;26(2):207-213. doi: 10.1177/1933719118818906. Epub 2018 Dec 12. PMID 30541396
- [Background] Kawamura K, Kawamura N, Hsueh AJ. Activation of dormant follicles: a new treatment for premature ovarian failure? Curr Opin Obstet Gynecol. 2016 Jun;28(3):217-22. doi: 10.1097/GCO.0000000000000268. PMID 27022685
- [Background] Nurden AT. Platelets, inflammation and tissue regeneration. Thromb Haemost. 2011 May;105 Suppl 1:S13-33. doi: 10.1160/THS10-11-0720. Epub 2011 Apr 11. PMID 21479340
- [Background] Gurtner GC, Werner S, Barrandon Y, Longaker MT. Wound repair and regeneration. Nature. 2008 May 15;453(7193):314-21. doi: 10.1038/nature07039. PMID 18480812
- [Background] Lacci KM, Dardik A. Platelet-rich plasma: support for its use in wound healing. Yale J Biol Med. 2010 Mar;83(1):1-9. PMID 20351977
- [Background] Sfakianoudis K, Simopoulou M, Nitsos N, Rapani A, Pantou A, Vaxevanoglou T, Kokkali G, Koutsilieris M, Pantos K. A Case Series on Platelet-Rich Plasma Revolutionary Management of Poor Responder Patients. Gynecol Obstet Invest. 2019;84(1):99-106. doi: 10.1159/000491697. Epub 2018 Aug 22. PMID 30134239
- [Background] Sills ES, Rickers NS, Li X, Palermo GD. First data on in vitro fertilization and blastocyst formation after intraovarian injection of calcium gluconate-activated autologous platelet rich plasma. Gynecol Endocrinol. 2018 Sep;34(9):756-760. doi: 10.1080/09513590.2018.1445219. Epub 2018 Feb 28. PMID 29486615
- [Background] Sills ES, Li X, Rickers NS, Wood SH, Palermo GD. Metabolic and neurobehavioral response following intraovarian administration of autologous activated platelet rich plasma: First qualitative data. Neuro Endocrinol Lett. 2019 Jan;39(6):427-433. PMID 30796792
- [Background] Sills ES, Rickers NS, Svid CS, Rickers JM, Wood SH. Normalized Ploidy Following 20 Consecutive Blastocysts with Chromosomal Error: Healthy 46, XY Pregnancy with IVF after Intraovarian Injection of Autologous Enriched Platelet-derived Growth Factors. Int J Mol Cell Med. 2019 Winter;8(1):84-90. doi: 10.22088/IJMCM.BUMS.8.1.84. Epub 2019 May 15. PMID 32195207
- [Background] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- See also: Ovarian rejuvenation and folliculogenesis reactivation in peri-menopausal women after autologous platelet-rich plasma treatment — https://sa1s3.patientpop.com/assets/docs/111052.pdf